CLINICAL TRIAL: NCT03765229
Title: Breaking Innate PD-1 Inhibitor (PD1i) Resistance Using Epigenetic Modifiers; Antitumor Efficacy and Correlative Analyses of Entinostat Plus Pembrolizumab in Non-Inflamed Metastatic Melanoma (MM)
Brief Title: An Exploratory Study of Pembrolizumab Plus Entinostat in Non-Inflamed Stage III/IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC1729
Record Dates: First submitted 2018-11-15; First posted 2018-12-05 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Melanoma
Keywords: PD-1
MeSH Terms: conditions — Melanoma | interventions — entinostat; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: Entinostat + Pembrolizumab (Experimental): Subjects in this trial will be administered entinostat, 5mg PO, once weekly (D1, D8, D15 of a 21-day cycle) starting on day 1 of study treatment. Pembrolizumab, 200 mg will be administered intravenously (IV) every 3 weeks and initiated at cycle 2 after the mandatory research tumor biopsy in the end of cycle 1, beginning of cycle 2 (day 21±2 days),. Combination therapy with both agents will continue if subject is receiving clinical benefit from therapy for up to 27 weeks (8 cycles of combination therapy or approximately 6 months). Study therapy will be discontinued for intolerable toxicity, disease progression or for other reasons at the discretion of the investigator.
  Interventions: Drug: Entinostat; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Entinostat — Oral drug 5 mg taken once weekly for up to nine 3-week (21 day) cycles. Take on an empty stomach i.e., at least 2 hours after a meal and at least 1 hour before the next meal. On days when entinostat is administered on the same day as pembrolizumab, entinostat should be taken before the pembrolizumab infusion.
Drug: Pembrolizumab — 200 mg IV starting on Day 22 (cycle 2, Day 1) given every 3 weeks for up to 8 cycles.
  Other Names: Keytruda

SUMMARY:
Cancers develop in two different ways. First, cancer cells can become invisible to the immune system by stop having proteins on their surface that are required for the immune system to recognize them. In this scenario, tumors do not attract any immune cells (e.g. white blood cells) whatsoever or they do not attract specialized white blood cells against cancer cells, called lymphocytes. White blood cells are the type of immune cells that attack foreign cells, such as cancer cells or normal cells infected with viruses or bacteria. Second, cancer cells can still grow side-to-side with white blood cells but are able to hide from them. As a result, the white blood cells cannot find and attack the cancer cells. Different types of cancers have different chance of having immune cells in the tumor. For example, the possibility that immune cells are within skin melanomas is almost 50% whereas the possibility in melanoma of the eye is only 10%.

As a result, the first goal of this study is to understand whether entinostat can make a melanoma tumor more visible to the immune system. To see whether entinostat makes tumor more visible to the immune system, participants will have a mandatory tumor biopsy 3 weeks after starting entinostat therapy. Tumor tissue collected before and after participating in this study will be compared to see if there are more immune cells in the tumor after receive entinostat. The second goal of the study is to see if giving a combination of entinostat and pembrolizumab can shrink melanoma tumors of patients who did not have immune cells in tumors prior to treatment. The study will determine how many subjects cancer has become better or not changed 6 months after subjects have started treatment on the study. We will also determine what type of side effects occur in subjects receiving entinostat and pembrolizumab to look at the safety of this combination.

The investigators will also look at any changes in the DNA of melanoma before the study begins. As a result of these changes in DNA, there are often see differences in the proteins that work to create other proteins. In addition, the study will look into how entinostat may make melanoma cells more visible to the immune system by comparing proteins in tumors before and after treatment. Finally, the study will see if this treatment changes the numbers and types of immune cells that are found in the blood by comparing blood at different time points while patients are on the study.

DETAILED DESCRIPTION:
This is an exploratory (n=10-12 evaluable patients), open-label, single-arm, phase II study in patients with 'non-inflamed' unresectable regional or distant metastatic melanomas irrespective of prior treatment with PD-1/PD-L1 pathway inhibitors. The primary endpoint is to assess the incidence of histopathologic conversion of non-inflamed melanomas from patients with metastatic melanoma to 'inflamed' melanoma following single-agent entinostat "priming" (entinostat monotherapy). More specifically, patients with metastatic melanomas that have no evidence of tumor-infiltrating or tumor-associated lymphocytes (TIL/TAL), based on standard hematoxylin and eosin (H&E) staining of representative tumor sections (non-inflamed melanomas) will receive weekly entinostat for 3 weeks in cycle 1 (entinostat monotherapy; 5mg PO, qwk on D1, D8, D15 of cycle 1; cycle length = 21 days). Mandatory tumor tissue biopsies will be performed in the end of cycle 1, beginning of cycle 2 (day 21±2 days), immediately before treatment with concurrent entinostat (once weekly × 3) and pembrolizumab (200 mg q3wks) in cycles 2-9 (see section 5.2.1 drug dosing schema). Correlative studies will be performed at baseline and in the end of cycle 1, beginning of cycle 2 (day 21±2 days) to assess whether: (a) 3 weeks of entinostat monotherapy converts TIL/TAL-absent melanomas to TIL/TAL-present by histopathologic (H&E stain) analysis, (b) 3 weeks of single-agent entinostat induces changes in gene expression profiling by assessing distinct signatures as defined by RNA-sequencing signatures (RNA-seq; 'immune-high', innate anti-PD-1 resistance, and epigenetic 1-3), (c) 3 weeks of single-agent entinostat induces changes in histone-accessible DNA by performing formaldehyde-assisted isolation of regulatory elements (FAIRE)4, (d) conversion of non-inflamed to inflamed melanomas by single-agent entinostat and/or antitumor response to the entinostat-pembrolizumab combination is associated with a baseline signature that consists of distinct somatic mutation gene profile, global histone modification profile in melanoma tissue or peripheral blood mononuclear cells (PBMC), and/or abundance of entinostat targets in melanoma cells (HDAC 1, 2, 3, and 11). Up to 12 evaluable patients will be treated with entinostat plus pembrolizumab for up to 27 weeks (approximately 6 months) based on clinical benefit. Patients who continue to have clinical benefit at 27 weeks may continue therapy with pembrolizumab or any other PD-1/PD-L1 inhibitor, as per standard of care.Secondary exploratory endpoints involve: (a) assessment of antitumor response of entinostat administered concurrently with pembrolizumab at week 10 (or earlier if patient progresses), based on response rate per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). (b) assessment of the progression-free survival (PFS) rate at 27 weeks (approximately 6 months) of the entinostat-pembrolizumab combination. (c) determine the safety of the entinostat-pembrolizumab combination in patients with metastatic melanoma per NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE). (d) assessment of other exploratory biomarkers in tumor tissue and peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent.
* Subject has provided informed consent and Health Insurance Portability and Accountability Act (HIPAA) prior to initiation of any study-specific activities/procedures.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
* Histologically confirmed metastatic (regional or distant) melanoma of any subtype (cutaneous, mucosal, ocular).
* American Joint Committee on Cancer (AJCC) stage unresectable III or stage IV disease that is measurable by RECIST v1.1 criteria.
* Must agree to undergo one on-treatment tumor biopsy on day 22 (±2 days) of the study. Subjects for whom fresh samples cannot be safely provided (e.g., inaccessible tumor for biopsy or has metastatic lung lesion(s) as the only site of metastatic disease) will not be eligible for study participation.
* Must have available archival tissue and subjects have consented to allow collection of archived tumor blocks from previous surgeries confirming or treating unresectable stage III or distant metastatic disease. If more than one archived tumor blocks are available, two blocks have to be analyzed for the presence of Tumor-infiltrating lymphocyte/Tumor-associated lymphocyte (TIL/TALS). Archived tumor tissues must fulfill the following criteria based on two representative Hematoxylin & Eosin (H&E)-stained tissue sections: (1) the tumor surface area must be at least 1cm (squared), (2) no more than 20% of necrosis, (3) the ratio of viable tumor cells to tumor-associated stroma should be at least 60/40, (4) if TILs are present based on H&E stained sections, they must be ≤ 1% of the total number of cells in the specimen; the amount of tissue should be ≥ 1 cm2.

The study pathologists must sign off on the eligibility of archived tumor blocks before study enrollment. If archival tissue is unavailable or insufficient, fresh biopsy should be performed to confirm unresectable stage III or distant metastatic disease.

* Previous treatment with immune checkpoint inhibitors and chemotherapies is allowed on condition that the last treatment is at least 28 days prior to first dose of entinostat. Previous treatment with targeted therapies (e.g. Mitogen-activated protein kinase inhibitors) is allowed on condition that the last treatment was administered at least 15 days prior to first dose of entinostat).
* Demonstrate adequate organ function as defined in the protocol table; all screening labs to be obtained within 21 days prior to entinostat treatment.

  *Note: Hematology and other lab parameters that are ≤ grade 2 but still meet criteria for study entry are allowed. Furthermore, changes in laboratory parameters during the study should not be considered Adverse events (AEs) unless they meet criteria for dose modification(s) of study medication outlined by the protocol in Section 5.3.1 and/or worsen from baseline during therapy.
* A female of childbearing potential must have a negative serum pregnancy test during screening and a negative urine pregnancy test within 3 days prior to receiving the first dose of study drug. If the screening serum test is done within 3 days prior to receiving the first dose of study drug, a urine test is not required. A female of childbearing potential must agree to use effective contraception during the study and for 120 days after the last dose of study drug. A female of non-childbearing potential defined as (by other than medical reasons):

  -≥45 years of age and has not had menses for >2 years,
* Amenorrheic for <2 years without a hysterectomy and oophorectomy and a follicle-stimulating hormone value in the postmenopausal range upon pre-study (screening) evaluation,
* Post hysterectomy, oophorectomy or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure; otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of entinostat,
* If male, agrees to use an adequate method of contraception starting with the first dose of study drug through 120 days after the last dose of entinostat,
* See section 5.6.2 for information on acceptable methods of contraception.
* Experienced resolution of toxic effect(s) of the most recent prior anti-cancer therapy to Grade ≤1 (except alopecia or neuropathy) by CTCAE v5.0. Exceptions are patients who may have developed autoimmune-type side effects that require permanent hormonal replacement from previous therapies.
* If the patient underwent major surgery or radiation therapy, these procedures must have occurred at least 15 days prior to the first dose of entinostat. In addition, patients must have recovered from the toxicity and/or complications from the intervention to Grade ≤1.
* Subjects must be willing and able to comply with study procedures based on the judgment of the investigator or protocol designee.

Exclusion Criteria:

All subjects meeting any of the exclusion criteria at baseline will be excluded from study.

* Is receiving systemic steroid therapy or any other form of immunosuppressive therapy for autoimmune side effects related to previous use of immunotherapies for melanoma. Exceptions include episodic (up to 7 days) use of systemic steroids for common conditions while on study treatment (e.g. Chronic obstructive pulmonary disease (COPD) exacerbation, poison ivy), use of corticosteroids as replacement doses for adrenal or pituitary insufficiency.
* Has a known history of tuberculosis (Bacillus Tuberculosis) or human immunodeficiency virus (HIV 1/2 antibodies).
* Hypersensitivity to pembrolizumab or any of its excipients. Allergy to benzamide or inactive components of entinostat.
* Has known history of biopsy-proven (non-infectious) pneumonitis that required systemic steroids, or any evidence of current pneumonitis.
* Conditions that would preclude adequate absorption of oral medications (malabsorption, significant nausea and vomiting, resection of >100-cm of proximal small bowel, resection of >200-cm of distant small bowel).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including but not limited to:

  i. Myocardial infarction or arterial thromboembolic events within 6 months prior to screening or severe or unstable angina, New York Heart Association (NYHA) Class III of IV disease, or a QT corrected for heart rate interval > 470 msec,

ii. Uncontrolled hypertension (>150/90 in more than 60% of recorded BP measurements taken on 5 or more separate occasions, within 3 weeks of the first dose of entinostat; at least 3 recorded measurements required on each occasion) or diabetes mellitus (HbA1c >9.0 within 15 days from first dose of entinostat),

iii. Active infection requiring systemic antibiotic therapy by the first day of entinostat treatment,

iv. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

* If female, is pregnant or breastfeeding, or, if male, expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBs Ag) are eligible. HBV DNA test must be performed in these patients prior to study treatment if known history of viral hepatitis. Patients positive for hepatitis C virus (HCV) antibody are eligible, only if polymerase chain reaction is negative for HCV RNA.
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live-attenuated vaccines and are not allowed.
* History of prior malignancy, with the exception of the following:

  * Non-melanoma skin cancers, non-invasive bladder cancer, and carcinoma in situ of the cervix,
  * Prior history of prostate cancer provided the patient is not undergoing active systemic treatment other than hormonal therapy and has documented prostate-specific antigen that is undetectable (<0.2ng/mL),
  * Papillary thyroid cancer, even if patients may have just completed thyroidectomy within the last 2 years, have not received adjuvant radioactive iodine therapy, and were only recently diagnosed with asymptomatic papillary thyroid cancer and their surgery is pending,
  * Chronic lymphocytic leukemia (CLL) provided patient has isolated lymphocytosis (Rai stage 0) and does not require systemic treatment [for "B" symptoms, Richter's transformation, lymphocyte doubling time (<6 months), lymphadenopathy or hepatosplenomegaly],
  * Lymphoma, hairy-cell leukemia, or myelodysplasia, provided that patient is not on active systemic treatment and is in complete remission, as evidenced by positron emission tomography/computerized tomography (PET/CT) scans and bone marrow biopsies for at least 3 months,
  * History of any other malignancy provided patient has completed therapy and is free of disease for ≥ 2 years. If patient had other malignancy within the last 2 years from which he, or she, may have been completely cured by surgery alone, he may be considered to be enrolled on condition that the risk of development of distant metastatic disease based on the most recent AJCC staging system is less than 30%.
* Has known active (i.e. previously untreated) parenchymal central nervous system (CNS) metastases that are symptomatic, and/or more than one lesion with the largest diameter being > 5-mm and/or require antiepileptic drugs or systemic corticosteroids for management of intracranial symptoms. Patients with carcinomatous meningitis are also excluded. Exceptions are:

  * Subjects with previously treated brain metastases provided they are stable (i.e. without evidence of progression by brain Magnetic Resonance Imaging (MRI) or head CT with IV contrast) for at least 2 weeks prior to the first dose of entinostat. Any neurologic symptoms must have returned to baseline, and have no evidence of new or enlarging brain metastases, and are not using ongoing systemic corticosteroids for management of intracranial symptoms for at least 7 days prior to first dose of entinostat,
  * Patients with active (i.e. not treated with stereotactic radiosurgery), single, asymptomatic, up to 5-mm in largest diameter brain metastases (measured either by brain MRI with IV contrast or head CT with IV contrast measuring within 2 weeks prior to the first dose of entinostat).
* Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of entinostat.
* Subject is receiving prohibited medications or treatments as listed in section 5.5 of the protocol that cannot be discontinued/replaced by an alternative therapy.
* Prior treatment with Histone/deacetylase inhibitor (HDACi) for their melanoma.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stergios Moschos, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were enrolled in the study between 03/22/2019-05/24/2022, at one cancer center in the United States. A total of 11 participants consented, were found eligible and started to study. During the screening period, 22 subjects were consented to and 11 subjects did not enroll in the study since 10 of them were deemed not eligible and 1 subject expired.
Period: Overall Study
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects signed the informed consent and started to study treatment.
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 58.36 [38 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Conversions of Non-inflamed to Inflamed Melanoma
Description: Number of subjects with conversion from non-inflamed Tumor-infiltrating lymphocyte / Tumor-associated lymphocyte (TIL/TAL) absent before treatment to TIL/TAL present after treatment was assessed by histopathologic analysis. Representative 5-micron thick formalin fixed paraffin embedded sections collected from baseline and on-treatment (entinostat-alone, day 21 of the trial) were stained with hematoxylin and eosin on day 21 (on-treatment biopsy).
Time Frame: 3 weeks after start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Number analyzed (Participants) | 10
Participants
  Tumor-infiltrating lymphocyte increased | 3
  Tumor-infiltrating lymphocyte not increased | 7

2. Secondary Outcome: Overall Response Rate
Description: Radiographic response will be measured by Response Evaluation Criteria In Solid Tumors (RECIST) Criteria for Complete Response (CR), disappearance of all target lesions or Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. The Overall Response rate will be the percentage of subjects with CR or PR at 9 weeks after the start of treatment.
Time Frame: 9 weeks
Population: Subjects started to the study treatment and response evaluation per RECIST was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Number analyzed (Participants) | 11
Participants
  Complete Response or Partial Response | 3
  Stable Disease or Progression | 8

3. Secondary Outcome: Progression-Free Survival
Description: Progression Free Survival is measured as the rate of patients who are progression-free from the date of enrollment on study to the date of documented progression per RECIST 1.1. criteria or death. Per RECIST 1.1, Progressive Disease (PD), is a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 6 months
Population: Subjects who started the study treatment and tumor response was evaluated, median follow-up time 14.3 (2.5-36.8) months.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Number analyzed (Participants) | 11
Participants
  Alive with no evidence of disease | 1
  Alive with disease | 3
  Died from disease | 7

4. Secondary Outcome: Number of Participant With Adverse Events During the Concurrent Pembrolizumab-entinostat Combination
Description: Type of AEs that occur in subjects enrolled who receive at least one dose of therapy will be reported based on the NCI Common Terminology Criteria for Adverse Events v5.0 (NCI-CTCAE v.5.0). The NCI-CTCAE is a descriptive terminology utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm: Entinostat + Pembrolizumab
Number analyzed (Participants) | 11
Participants
  fatigue | 11
  nausea | 6
  vomiting | 3
  diarrhea | 7
  anorexia | 3
  musculoskeletal pain | 5
  cytopenia | 2
  anemia | 8

ADVERSE EVENTS:
Time Frame: Up to 90 days.
Description: Adverse events were collected from day one of the study drug administration to 30 days after completion of treatment. Any hospital admission was considered as a serious adverse event.
Groups:
- Single Arm: Entinostat + Pembrolizumab: Subjects in this trial will receive entinostat and pembrolizumab.
Arm/Group | Single Arm: Entinostat + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 7/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Entinostat + Pembrolizumab (N=11)
Anemia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (Gastrointestinal disorders) | 1
fatigue (General disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Musculoskeletal and connective tissue disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Hallucinations (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hematoma (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm: Entinostat + Pembrolizumab (N=11)
Anemia (Blood and lymphatic system disorders) | 8
Eosinophilia (Blood and lymphatic system disorders) | 2
Atrial fibrillation (Cardiac disorders) | 2
Palpitation (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Hearing impaired (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Blurred vision (Eye disorders) | 2
Dry eye (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Edema limbs (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 11
Fever (General disorders) | 2
Malaise (General disorders) | 1
Pain (General disorders) | 3
Hepatic pain (Hepatobiliary disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Bruising (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 5
Creatinine increased (Investigations) | 6
Investigations - Other, specify (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 11
Neutrophil count decreased (Investigations) | 5
Platelet count decreased (Investigations) | 6
Serum amylase increased (Investigations) | 1
Thyroid stimulating hormone increased (Investigations) | 2
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Obesity (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Memory impairment (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Radiculitis (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 5
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Hematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 6
Hypotension (Vascular disorders) | 2
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03765229/Prot_SAP_000.pdf